CLINICAL TRIAL: NCT03421756
Title: A Pilot Study Evaluating the Efficacy of Non-Myeloablative Matched Related Donor Peripheral Blood Stem Cell Transplant in Patients With Severe Sickle Cell Disease
Brief Title: Stem Cell Transplant in Patients With Severe Sickle Cell Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Trial terminated due to low rate of enrollment
Sponsor: Kathleen Dorritie (Other)
Responsible Party: Sponsor-Investigator, Kathleen Dorritie, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 17-097
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Alemtuzumab; Whole-Body Irradiation; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non Myeloablative regimen (Alemtuzumab) (Experimental): Sickle cell patient receives sibling donor peripheral blood stem cell transplant with non-myeloablative pre-transplant conditioning.
  Interventions: Drug: Alemtuzumab; Radiation: Total Body Irradiation; Drug: Sirolimus

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab is a non-myeloablative pre-transplant conditioning regimen. Non-myeloablative therapy uses doses of chemotherapy and radiation to weaken (but not destroy) the patients bone marrow and immune system, while still allowing their body will accept the donor's stem cells. Alemtuzumab will be given 7 days prior to stem cell infusion at 0.03 mg/kg IV, 6 days prior to stem cell infusion at 0.1 mg/kg IV, and 5 thru 3 days prior to stem cell infusion at 0.3 mg/kg IV.
Radiation: Total Body Irradiation — 300 cGy will be administered in a single fraction on Day - 2. TBI is used commonly as part of pre-transplant conditioning in a variety of settings.
  Other Names: TBI
Drug: Sirolimus — Sirolimus will be used for the prevention of graft-verus-host disease and will begin on Day - 1.
  Other Names: Rapammune

SUMMARY:
This is a prospective pilot study of matched-related donor allogeneic stem cell transplantation in adults with severe sickle cell disease using a matched-sibling PBSC graft with a non-myeloablative conditioning regimen (Alemtuzumab).

DETAILED DESCRIPTION:
Stem cell transplantation recipients will be given Alemtuzumab, which is a non-myeloablative pre-transplant conditioning regimen. This non-myeloablative therapy uses doses of chemotherapy and radiation to weaken (but not destroy) the patients bone marrow and immune system, while still allowing their body to accept the donor's stem cells. Alemtuzumab will be given 7 days prior to stem cell infusion at 0.03 mg/kg IV, 6 days prior to stem cell infusion at 0.1 mg/kg IV, and 5 thru 3 days prior to stem cell infusion at 0.3 mg/kg IV.

ELIGIBILITY:
Inclusion Criteria:

* Patient selection

  1. Age > 18 years
  2. Patients with Hb SS, Hb SC, Hb Sβ0 genotype
  3. Presence of at least 1 of the following manifestations:

     1. History of clinically significant neurologic event defined as stroke or any neurological deficit lasting > 24 hours.
     2. History of two or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures
     3. Three or more pain crises per year in the 2-year period preceding referral (required intravenous pain management in the outpatient or inpatient hospital setting).

        This may include painful episodes related to priapism, osteonecrosis or any sickle-related complication.
     4. An echocardiographic finding of the tricuspid valve regurgitant jet (TRJ) velocity ≥ 2.7 m/sec.
     5. History of osteonecrosis or avascular necrosis of ≥ 2 joints
     6. Administration of regular RBC transfusion therapy, defined as receiving 8 or more transfusions per year for > 1 year to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and acute chest syndrome)
     7. History of RBC allo-immunization but without detectable allo-antibodies.
     8. Evidence of sickle hepatopathy or iron overload in patients who received ≥ 8 packed RBC transfusions for ≥ 1 year or have received ≥ 20 cumulative packed RBC transfusions. These patients will undergo MRI of the liver to estimate liver iron content.
     9. Patients with hepatic iron content of ≤ 7 mg Fe/ gm of liver will be included ii. Patients with hepatic iron content of ≥ 7 mg Fe/ gm of liver will undergo biopsy to look for absence of histological findings suggestive of cirrhosis, fibrosis and active hepatitis

     h. Sickle nephropathy defined as Cr ≥ 1.5 times the ULN or biopsy proven i.Reversible SCD complication not ameliorated by hydroxyurea: i.Two or more vaso-occlusive crises requiring hospitalizations ii. Any episode of ACS while on hydroxyurea
  4. Adequate physical function as measured by all of the following:

     1. Karnofsky performance score > or equal to 70
     2. Cardiac function: Left ventricular ejection fraction (LVEF) > 40%; or LV shortening fraction > 26% by cardiac echocardiogram or by MUGA scan.
     3. Pulmonary function: Pulse oximetry with a baseline O2 saturation of > 85%, DLCO > 40% (corrected for hemoglobin).
     4. Renal function: Serum creatinine ≤ 1.5 x the upper limit of normal for age as per local laboratory and 24 hour urine creatinine clearance >70 mL/min/1.73 m2; or GFR > 70 mL/min/1.73 m2 by radionuclide GFR unless reason for transplant is sickle nephropathy
     5. Hepatic function:

     i. Serum conjugated (direct) bilirubin < 2x upper limit of normal for age as per local laboratory; ii. ALT and AST < 5 times upper limit of normal. iii. Patients with hyperbilirubinemia because of hyper hemolysis, or who experience a sudden, profound change in the serum hemoglobin after a RBC transfusion are not excluded.
  5. The HLA matched related donor must be willing to donate and must meet our institutional guidelines to donate peripheral blood stem cells
  6. Absence of donor specific HLA antibodies.
  7. Absence of clinical or radiographic evidence of neurologic event within 6 months prior to proceeding with transplantation.

     1. Cerebral MRI/MRA within 6 months prior to initiation of transplant conditioning.
     2. If patient has a neurologic event such as stroke or transient ischemic attack during recruitment process, patient will be deferred for 6 months before reconsideration.

Donor selection

1. Siblings who are ≥18 years and capable and willing to donate PBSC
2. Sibling donors are HLA-matched. HLA-A, B, C, and DRB1 match based on high-resolution typing
3. All sibling donors MUST meet institutional criteria for donation.
4. Donors with sickle cell trait (Hb AS) are permitted.
5. Donors with ABO minor incompatibility are permitted

Exclusion Criteria:

Patient selection

1. Uncontrolled bacterial, viral or fungal infection in the 6 weeks before enrollment.
2. Seropositivity for HIV.
3. Previous stem cell transplantation.
4. Participation in a clinical trial in which the patient received an investigational drug or device
5. A history of substance abuse as defined by version IV of the Diagnostic & Statistical Manual of Mental Disorders (DSM IV).
6. Demonstrated lack of compliance with prior medical care as determined by referring physician.
7. Pregnant or breast-feeding females.
8. Unwillingness to use approved contraception method from time of conditioning regimen and 4 months after discontinuation of all immunosuppressive medications.

Donor selection A. Inclusion Criteria

1. Siblings who are ≥18 years and capable and willing to donate PBSC
2. Sibling donors are HLA-matched. HLA-A, B, C, and DRB1 match based on high-resolution typing
3. All sibling donors MUST meet institutional criteria for donation.
4. Donors with sickle cell trait (Hb AS) are permitted.
5. Donors with ABO minor incompatibility are permitted

B. Exclusion Criteria

1. Donors with hemoglobinopathies: Hb SS, Hb SC, Hb Sβ0 and all other unstable hemoglobins
2. Presence of anti-donor HLA antibodies in the recipient
3. Donors with major ABO incompatibility are permitted
4. Donors who are HIV-1, HIV-2, HTLV-1, HTLV-2 seropositive or with active hepatitis B or hepatitis C virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Treatment Success | up to 1 year after HSCT
  Evaluating reversal of Hb S % to that of the donor's phenotype, in recipients of HLA matched-sibling peripheral blood - hematopoietic stem cell transplantation (HSCT) with NMA conditioning regimen. Testing for treatment success will include Hb Electrophoresis. Recipients with donors AA should have nearly 0% Hb S. Recipients with donors AS should have similar Hb S % (approximately < 60%) as the donor. The proportion of patients experiencing treatment success, will be calculated with a 90% exact confidence interval.

SECONDARY OUTCOMES:
Engraftment | up to 1 year after HSCT
  To estimate the probability of engraftment, using absolute neutrophil count and platelets along with chimerism analysis after HSCT. This will by evaluated by: 1) Time to ANC of >500/uL on the first of three consecutive days. 2) Time to platelet count >50,000/µL for 3 days without transfusion. 3) Peripheral blood chimerism analysis of whole blood and CD3-lineage will be performed on or around day +30, +90, +180, and +360. 4) Additional peripheral blood chimerism studies may be performed as clinically indicated. The statistical analysis plan will be calculated with a 90% exact confidence interval.
Probability of developing acute GVHD after HSCT. | up to 100 days after HSCT
  Acute GVHD will be diagnosed and graded using the clinical and laboratory criteria in Appendix A of the protocol. During the inpatient stay, clinical evaluations will occur daily. During the outpatient stay, each patient should be evaluated at least every other week until they are discharged from the transplant clinic. Subsequent evaluations will occur at roughly Days +30, +60, +90 and until +100 days. Clinical evaluations will be performed and grade will be assigned at the time of diagnosis by an attending physician. The decision to initiate GVHD therapy will be made by the attending physician. The statistical analysis plan will be calculated with a 90% exact confidence interval.
Probability of developing chronic GVHD after HSCT. | up to 2 years after HSCT
  Chronic GVHD will be diagnosed using NIH criteria outlined in Appendix B of the protocol. b. Evaluation will be conducted by BMT team at day +100, +360 and yearly up to 2 years after HCT. The patient's sickle cell physician will conduct clinical assessments between these time points as required per institutional guidelines. This will be evaluate by: 1) The occurrence of chronic GHVD meeting NIH criteria and requiring systemic pharmacological immunosuppression 2) The use of additional immune suppressive agents other than first line therapy 3) Time to completion of prednisone, if required for treatment of acute GVHD 4) Time to completion of all immunosuppression 5) Requirement for immunosuppression at 1 year and 2 years after transplant. The statistical analysis plan will be calculated with a 90% exact confidence interval.
Graft failure or Relapse | up to 2 years after HSCT
  Relapse is defined by the presence of recipient's Hb SS on electrophoresis. Testing for recurrent disease will include Hb electrophoresis to determine recipient vs. donor Hb-type and peripheral blood chimerism to document loss of donor cell engraftment. Endpoints will include: time to relapse and status of compliance with immunosuppressive therapy. Primary graft failure defined as the absence of donor cells assessed by peripheral blood chimerism assays, by any lineage, on or after day +30. Secondary graft failure defined as the presence of < 20% donor cells by peripheral blood chimerism assays in a patient with prior evidence of ≥ 20% of donor cells. The analysis plan for graft failure or relapse will be calculated with a 90% exact confidence interval.
Discontinuation of Immunosuppressive therapy | up to 2 years after HSCT
  The time (in days) it takes to taper immunosuppressive therapy will be measured. Tapering will begin once 50% donor CD3 chimerism is achieved. To estimate the time to discontinuation of immunosuppressive therapy. The product-limit (Kaplan-Meier) estimate of the distribution of time to discontinuation will be calculated with a 90% confidence region. In an exploratory analysis, proportional hazards (Cox) regression will be applied to identify potential predictors of time to discontinuation.
Sickle cell disease related organ damage | up to 2 years after HSCT
  Cardiac function, pulmonary function, renal function, cerebrovascular function will be measured. We will measure and record BNP, left atrial diameter and the tricuspid regurgitant velocity, noted on transthoracic echocardiogram, (TTE) as a marker of improvement at an outpatient cardiology follow-up visit. We will measure and record a 6-minute walking distance test and pulmonary function test variables to include: FEV1, FVC, TLC, RV, DLCO, and O2 saturation at an outpatient pulmonology follow-up visit.We will measure and record the urine-albumin creatinine ratio as a measure of micro-/macro-albuminuria and 24-hr urine proteinat an outpatient nephrology follow-up visit.We will obtain a brain MRI at an outpatient neurology follow-up visit. All evaluations will take place at baseline, Day +365, and Day +720.
Lymphocyte subsets | up to 2 years after HSCT
  To evaluate lymphocyte subsets. This analysis will be descriptive.
Changes in monthly transfusions after HSCT | up to 2 years after HSCT
  We will monitor the number of transfusions required on a monthly basis pre- and post-HSCT Patient's monthly transfusions will be recorded starting 3 months pre-HSCT. Patient's monthly transfusions will be recorded post-HSCT at the following time points: Days +30, +60, +90, +180, +365, +720. To evaluate changes in monthly transfusion dependence after HSCT in patients, will be modeled using mixed effects regression.
Changes in the annual frequency of SCD-related hospitalization after | up to 2 years after HSCT
  The patients frequency of hospital stays will be measured compared to prior HSCT. Number of hospitalizations per year post-HSCT will be recorded at Days 0, +365 and +720. A mixed effects Poisson regression model will compare the patients' frequency of hospitalization three years pre-transplant to post-transplant.
Quality of life measures | up to 2 years after HSCT
  Quality of life will be measured utilizing validated tools as well as new tools specific for sickle cell disease including the questionnaires: SF-36, Adult Sickle Cell Quality of life Measurement Information System (ASCQ-Me), Pittsburgh Sleep Quality Index, Generalized Anxiety Disorder-7, Brief Pain Inventory, and Painimation. To evaluate improvement in quality of life measures after HSCT. The recommended summary indices for the quality of life instruments will be calculated and their change over time by mixed effects linear models.
Transplant-related mortality | up to 2 years after HSCT
  TRM is defined as mortality in any patient for whom there has not been a diagnosis of relapse.To estimate transplant-related mortality: The product-limit (Kaplan-Meier) estimate of the distribution of time to discontinuation will be calculated with a 90% confidence region. In an exploratory analysis, proportional hazards (Cox) regression will be applied to identify potential predictors of time to discontinuation.
Opioid independence | up to 2 years after HSCT
  We will monitor the narcotic use in all recipients. At our institution, opioid adjustments are made by our SCD physicians who will be caring for these patients both pre- and post-transplant.
  Information on weekly narcotic use will be obtained and will be converted to the oral morphine equivalent (OME) dose for data collection. This will be done for the one week duration immediately prior to the following time points: Days 0, +30, +60, +90, +180, +365, +720.
MDC, whole blood and CD3 Lineage | up to 1 year after HSCT
  To estimate the probability of MDC, whole blood and CD3-lineage at 1 year.The statistical analysis plan will be calculated with a 90% exact confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Dorritie, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No